CLINICAL TRIAL: NCT06566183
Title: ISCHEMIA-LVD: International Study of Comparative Health Effectiveness With Medical and Invasive Approaches-Left Ventricular Dysfunction Trial
Brief Title: International Study of Comparative Health Effectiveness With Medical and Invasive Approaches-Left Ventricular Dysfunction Trial
Acronym: ISCHEMIA-LVD
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pending
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Coronary Artery Disease; Cognitive Impairment; Heart Failure
Keywords: Coronary Artery Disease; Heart Failure; Ejection Fraction
MeSH Terms: conditions — Coronary Artery Disease; Cognitive Dysfunction; Heart Failure | interventions — Coronary Artery Bypass; Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GDMT (Experimental): Participants with multivessel coronary artery disease (CAD) and heart failure with reduced ejection fraction (HFrEF) who are assigned to receive GDMT.
  Interventions: Procedure: Guideline-directed medical therapy (GDMT)
- CABG (Experimental): Participants with multivessel coronary artery disease (CAD) and heart failure with reduced ejection fraction (HFrEF) who are assigned to receive CABG.
  Interventions: Procedure: Coronary artery bypass grafting (CABG)
- PCI (Experimental): Participants with multivessel coronary artery disease (CAD) and heart failure with reduced ejection fraction (HFrEF) who are assigned to receive PCI.
  Interventions: Procedure: Percutaneous coronary intervention (PCI).

INTERVENTIONS:
Procedure: Guideline-directed medical therapy (GDMT) — Participants receive guideline-directed medical therapy (GDMT).
  Arms: GDMT
Procedure: Coronary artery bypass grafting (CABG) — Participants receive coronary artery bypass grafting (CABG).
  Arms: CABG
Procedure: Percutaneous coronary intervention (PCI). — Participants receive percutaneous coronary intervention (PCI).
  Arms: PCI

SUMMARY:
The ISCHEMIA-HF trial will randomize participants with multivessel coronary artery disease (CAD) with ejection fraction (EF) ≤40% in a 1:2:2 fashion to guideline-directed medical therapy (GDMT):coronary artery bypass grafting (CABG):percutaneous coronary intervention (PCI).

ELIGIBILITY:
Inclusion Criteria:

* Left ventricular ejection fraction (LVEF) ≤ 40% within prior 6 months (any local measurement, made within the past 6 months using echocardiography, multigated acquisition (MUGA), computed tomography (CT) scanning, magnetic resonance imaging (MRI), or ventricular angiography is acceptable, provided no subsequent measurement above 40%)
* Participants with multivessel CAD (defined as severe 3 vessel disease or 2 vessel disease including left anterior descending (LAD) artery disease) on coronary CT angiography (CCTA) or invasive coronary angiography
* CAD amenable to either PCI or CABG as determined by the local heart team
* Participant is willing to comply with all aspects of the protocol, including adherence to the assigned strategy, medical therapy and follow-up visits
* Participant is able and willing to give written informed consent

Exclusion Criteria:

* Decompensated heart failure or cardiogenic shock in the past 48 hours prior to randomization
* Concomitant significant valvular heart disease requiring surgery
* Prior cardiac surgery
* Dementia with loss of capacity to consent (clinically evident or previously diagnosed)
* Stroke within the previous 6 months or spontaneous intracranial hemorrhage at any time
* History of noncompliance with medical therapy
* Life expectancy less than the duration of the trial due to non-cardiovascular comorbidity
* Pregnancy (known to be pregnant; to be confirmed before randomization, if applicable)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Composite Cognitive Score | Month 12
  A composite score of various cognitive measures. Note that the total score range, calculation and interpretation to be updated upon submission of study protocol/materials to NYU Grossman School of Medicine IRB.
Kansas City Cardiomyopathy Questionnaire (KCCQ) Score | Month 12
  The KCCQ is an 8-item assessment of heart failure (HF)-related health status. The raw score is calculated using the response to each item; the total score transforms the raw score to a standardized score scaled from 0 to 100 and summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent.
Composite Number of: Death, Nonfatal Myocardial infarction (MI), Stroke, and Hospitalization for HF | Month 12
  Composite calculation of the number participants who experience death, nonfatal MI, stroke, or hospitalization for HF in each arm.

SECONDARY OUTCOMES:
Composite Number of: Mild Cognitive Impairment (MCI), Probable Dementia or Persistent Disability | Month 12
  Composite calculation of the number of participants with MCI, probable dementia or persistent disability in each arm.
Composite Number of: Death or Hospitalization for HF | Month 12
  Composite calculation of the number of participants who die or are hospitalized for HF in each arm.
Composite Number of: Death or Hospitalization for Cardiovascular (CV) Cause | Month 12
  Composite calculation of the number of participants who die or are hospitalized due to CV-related causes in each arm.
Seattle Angina Questionnaire (SAQ) Physical Limitations and Quality of Life Domain Score | Month 12
  The SAQ Physical Limitations and Quality of Life domain comprises 2 items of the SAQ corresponding with angina-related physical limitations and quality of life (QOL). The raw score is calculated using the response to each item; the total score transforms the raw score to a standardized score scaled from 0 to 100 and summarized in 25-point ranges where: 0 to 24 represents poor health status, 25 to 49 represents fair status, 50 to 74 represents good status, and 75 to 100 represents excellent status.
Self-Care of Heart Failure Index (SCHFI) | Month 12
  The SCHFI is a 39-item questionnaire assessing HF patients' performance of self-care activities related to HF, including how often they complete self-care, how likely they are to perform certain activities, and how confident they feel in performing the activities. Each item is rated on a scale from 1-5; the total score is the sum of responses and ranges from 39-195. Higher scores indicate greater overall performance of self-care activities related to HF.

CONTACTS AND LOCATIONS:
Overall Officials: S. Bangalore, MD, Principal Investigator — NYU Langone Health
Locations (6):
- NYU Langone Health, New York, New York, United States
- International Study Site, International Study Site, Brazil
- International Study Site, International Study Site, India
- International Study Site, International Study Site, Mexico
- International Study Site, International Study Site, Poland
- International Study Site, International Study Site, South Korea

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Sripal.bangalore@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Sripal.bangalore@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.